CLINICAL TRIAL: NCT01580774
Title: Effect of Post-discharge Phone Calls on Patient Outcomes for General Internal Medicine Patients Discharged From a Teaching Hospital.
Brief Title: Effect of Post-discharge Phone Calls on Patient Outcomes
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Christine Soong, Assistant Professor, Mount Sinai Hospital, Canada
Other Study IDs: MSHCANADA-CSCB
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Transition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post-discharge phone call: All patients in this group will receive a phone call within 72-hours of being discharged from hospital.
- Usual care (no phone call)

SUMMARY:
The purpose of this study is to determine whether a post-discharge telephone call to general medical patients discharged home will improve quality of care and adherence, and reduce hospital readmission.

DETAILED DESCRIPTION:
Currently, discharge from hospital in many institutions is a confusing process for patients filled with uncertainty and potential for harm. For instance, 1 in 5 discharges results in a post discharge adverse event, many of which are related to medication errors. These may lead to serious harm and possibly require readmission to hospital. Telephone follow-up calls after discharge has been studied in small single-center trials and as a part of a coordinated, multi-layered discharge process but its direct effectiveness is not known. Understanding the impact of this simple intervention on patient outcomes is an important step towards improving patients' discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Admission to internal medicine ward
* Discharged to home
* Must have telephone access

Exclusion Criteria:

* Discharged to care facility
* Lack of telephone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is patients admitted to a general internal medicine ward.
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Care Transition Measure-3 score (CTM-3) | 30-days post discharge

SECONDARY OUTCOMES:
Hospital readmission | 30-day post discharge
Emergency department visit | 30-days post discharge
Patient satisfaction | 30-days post discharge
Treatment plan adherence | 30-days post discharge
Outpatient provider follow-up rates | 30-days post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christine Soong, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Soong C, Kurabi B, Wells D, Caines L, Morgan MW, Ramsden R, Bell CM. Do post discharge phone calls improve care transitions? A cluster-randomized trial. PLoS One. 2014 Nov 11;9(11):e112230. doi: 10.1371/journal.pone.0112230. eCollection 2014. PMID 25386678